CLINICAL TRIAL: NCT01639313
Title: Is Arterial Pulse Contour Analysis Using Nexfin a New Option in the Non-invasive Measurement of Cardiac Output? - A Pilot Study
Brief Title: Comparison of Nexfin Pulse Contour Analysis and Cardiac Magnetic Resonance Imaging for the Measurement of Cardiac Output
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: PCA_CMR_MA
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A growing interest in monitoring cardiac output (CO) non-invasively has emerged, however its determination has been difficult using the standard approaches. The aim of the study is to evaluate the accuracy and precision of pulse contour analysis (PCA) as compared to cardiac magnetic resonance imaging (CMR).

ELIGIBILITY:
Inclusion Criteria:

* indication for CMR

Exclusion Criteria:

* contraindication for CMR
* claustrophobia
* no consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodynamically stable patients undergoing CMR
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany